CLINICAL TRIAL: NCT03248947
Title: Buprenorphine Physician-Pharmacist Collaboration in the Management of Patients With Opioid Use Disorder: Clinical Trials Network 0075
Brief Title: Buprenorphine Physician-Pharmacist Collaboration in the Management of Patients With Opioid Use Disorder: CTN 0075
Acronym: Pharm-OUD-Care
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083544; UG1DA040317 (NIH)
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; Medication-assisted treatment; Buprenorphine treatment; Collaborative care model
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pharmacy opioid use disorder care (Other): A single-arm study to evaluate the feasibility and acceptability of transitioning office-based buprenorphine treatment of adult patients with opioid use disorder from physicians to pharmacists.
  Interventions: Drug: buprenorphine/naloxone; Other: Pharmacist-administered buprenorphine/naloxone maintenance care

INTERVENTIONS:
Drug: buprenorphine/naloxone — To relieve opioid withdrawal symptoms and craving, buprenorphine/naloxone will be prescribed by the study-physician and dispensed by the study-pharmacist on a monthly basis. The median expected dose is 16 mg daily, though adjustment by the study physician may be needed due to increased withdrawal and craving from previous study visits. Medication will be provided in the form of a sublingual film.
Other: Pharmacist-administered buprenorphine/naloxone maintenance care — Following buprenorphine/naloxone induction/stabilization with the physician, participants with opioid use disorder will be transferred to the care of pharmacists for the maintenance phase of treatment. Maintenance visits will occur monthly with the pharmacist at the pharmacy location for six months. Buprenorphine/naloxone will be dispensed by the pharmacist at the monthly study visits following participant assessment, communication with the physician, and prescription form the physician.

SUMMARY:
This pilot study examines the feasibility and acceptability of transitioning office-based buprenorphine treatment of opioid use disorder from physicians to pharmacists. Results from this study will inform the development of a future multi-site randomized clinical trial.

DETAILED DESCRIPTION:
The overall objective of this study is to explore the feasibility of transitioning the care of adult patients with opioid use disorder (OUD) who receive office-based buprenorphine treatment (OBBT) from physicians to pharmacists. Physicians will induce buprenorphine treatment and complete the stabilization phase before referring patients to pharmacists for the management of monthly maintenance visits. This study will assess the feasibility and acceptability of a collaborative care model between physician and pharmacist by measuring recruitment rate, treatment retention rate, treatment compliance rate, and participants' substance use. Other assessments measured will include treatment fidelity, participant, physician, and pharmacist satisfaction with OUD care, participant safety, and the pharmacists' use of electronic health records and the Prescription Drug Monitoring Program.

ELIGIBILITY:
Inclusion Criteria:

* Be adults aged 18 years or older.
* If female, use adequate birth control methods.
* Meet DSM-5 criteria for past-year OUD and have completed buprenorphine induction for OUD.
* Have expressed the intention to receive maintenance (≥6 months) buprenorphine treatment.
* Be willing to receive pharmacist administered buprenorphine maintenance treatment
* Be willing and able to provide written informed consent and HIPAA authorization.
* Be able to read and communicate in English.
* Be able to comply with buprenorphine treatment policies.

Exclusion Criteria:

* Have a serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make study participation hazardous to the participant, compromise study findings, or prevent the participant from completing the study.
* Have known allergy or hypersensitivity to buprenorphine, naloxone, or other components of the buprenorphine/naloxone formulation.
* Have aspartate aminotransferase (AST) or alanine aminotransferase (ALT) liver enzymes greater than 5 times the upper limit of normal on screening phlebotomy performed within 60 days prior to the date of the last stabilization visit.
* Have chronic pain requiring ongoing pain management with opioid analgesics.
* Pending legal action or other reasons that might prevent an individual from completing the study (i.e., unable to complete 6 months of pharmacy-based OUD management).
* Pregnant or breastfeeding at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzy Wu, Sc.D., Principal Investigator — Professor; Paolo Mannelli, M.D., Principal Investigator — Associate Professor
Locations (6):
- United States (6):
  - Duke Outpatient Clinic, Durham, North Carolina
  - Josefs Pharmacy, Durham, North Carolina
  - Changes by Choice, Durham, North Carolina
  - Clinic Pharmacy, Durham, North Carolina
  - Carolina Performance, Raleigh, North Carolina
  - Health Park Pharmacy, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu LT, John WS, Ghitza UE, Wahle A, Matthews AG, Lewis M, Hart B, Hubbard Z, Bowlby LA, Greenblatt LH, Mannelli P; Pharm-OUD-Care Collaborative Investigators. Buprenorphine physician-pharmacist collaboration in the management of patients with opioid use disorder: results from a multisite study of the National Drug Abuse Treatment Clinical Trials Network. Addiction. 2021 Jul;116(7):1805-1816. doi: 10.1111/add.15353. Epub 2021 Jan 11. PMID 33428284

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacist-administered Buprenorphine Maintenance Care: Following buprenorphine/naloxone induction/stabilization with the physician, participants with opioid use disorder will be transferred to the care of pharmacists for the maintenance phase of treatment. Maintenance visits will occur monthly with the pharmacist at the pharmacy location for six months. Buprenorphine/naloxone will be dispensed by the pharmacist at the monthly study visits following participant assessment, communication with the physician, and prescription form the physician.
Period: Overall Study
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Started | 71
Completed | 63
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 61
  More than one race | 0
  Unknown or Not Reported | 1
Opioid positive UDS at screening [Count of Participants; unit: Participants] — UDS = urine drug screening
  Participants | 6

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Measured by a composite of the number of participants with opioid use disorder recruited (i.e., signed the informed consent form) per month, and by site and the average monthly rate of participants enrolled among potential participants who were screened.
Time Frame: Up to six months
Measure: Count of Participants; unit: Participants
Groups:
- Pre-screened Participants: Potential study participants who were approached by research staff to assess basic study eligibility and interest in study participation.
- Consented Participants: Participants who signed the study informed consent form and then underwent screening to determine study eligibility.
Arm/Group | Pre-screened Participants | Consented Participants
Number analyzed (Participants) | 92 | 76
Participants
  Pre-screened participants consented | 76 | NA — Row data only applies to pre-screened participants.
  Consented participants enrolled into study | NA — Row data only applies to consented participants. | 71

2. Primary Outcome: Treatment Retention
Description: Number of scheduled visits completed.
Time Frame: Up to six months
Population: The number of expected study visits for each participant is 6, based on 1 visit per month for the 6 months of the study arm. The overall number of expected study visits for all participants is 426, based on 6 visits per participant multiplied by 71 participants in the study arm.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Number analyzed (Visits) | 426
Visits | 406

3. Primary Outcome: Number of Participants With Opioid and Other Substance Use
Description: Measured via a composite of urine drug screen (UDS) and self-report via Timeline Follow-Back over 30 days.
Time Frame: Up to six months
Population: Missing UDS imputed as positive
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Participants
  Positive opioid UDS at month 6 | 10
  Positive other substance UDS at month 6 | 38
  Self-reported opioid use at month 6 | 10

4. Primary Outcome: Number of Medication-Compliant Months Across All Participants
Description: Medication compliance is defined as taking any of the dispensed medication during the past month as measured by pill count/dose reconciliation at each study visit. Medication compliance is calculated as the percentage of compliant months out of the overall number of expected study months.
Time Frame: Up to six months
Measure: Count of Units; unit: Months
Units Other Than Participants: Months
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Number analyzed (Months) | 426
Months | 406

5. Secondary Outcome: Treatment Fidelity
Description: Number of monitored study visits with physicians and pharmacists showing 80% adherence or higher to study specific tasks and responsibilities. Adherence will be calculated as the number of items completed on the Buprenorphine Visit Checklist divided by the sum of the number of complete and incomplete items.
Time Frame: Up to six months
Population: A total of 142 study visits were monitored for adherence to study tasks and responsibilities via completion of the Buprenorphine Visit Checklist. The percentage of monitored study visits with 80% adherence out of the total number of monitored study visits was calculated.
Measure: Count of Units; unit: Monitored study visits
Units Other Than Participants: Monitored study visits
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Number analyzed (Monitored study visits) | 142
Monitored study visits | 142

6. Secondary Outcome: Treatment Satisfaction
Description: Indicators of satisfaction with treatment delivery measured by participants, pharmacists, and physicians using the Treatment Satisfaction Scale after each study visit. A score of 5=very satisfied, 4=satisfied, 3=neither satisfied or dissatisfied, 2=dissatisfied, and 1=very dissatisfied.
Time Frame: Up to six months
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Study Physicians and Pharmacists: Comprised of the physicians (n=6) and pharmacists (n=6) who participated in the study.
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care | Study Physicians and Pharmacists
Number analyzed (Participants) | 63 | 12
Participants
  Overall satisfaction with experience in study: Very Satisfied | 59 | 12
  Overall satisfaction with experience in study: Satisfied | 3 | 0
  Overall satisfaction with experience in study: Neither Satisfied or Dissatisfied | 0 | 0
  Overall satisfaction with experience in study: Dissatisfied | 1 | 0
  Overall satisfaction with experience in study: Very Dissatisfied | 0 | 0
  Overall satisfaction with quality of study treatmt: Very Satisfied | 57 | 11
  Overall satisfaction with quality of study treatmt: Satisfied | 5 | 1
  Overall satisfaction with quality of study treatmt: Neither Satisfied or Dissatisfied | 0 | 0
  Overall satisfaction with quality of study treatmt: Dissatisfied | 1 | 0
  Overall satisfaction with quality of study treatmt: Very Dissatisfied | 0 | 0

7. Secondary Outcome: Participant Safety
Description: A composite of self-report and medical record abstraction to measure any fatal or non-fatal opioid overdose and any opioid or other substance-related emergency department visit or hospitalization.
Time Frame: Up to six months
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Participants
  Overdoses | 0
  Substance-related ED visits | 1
  Substance-related hospitalizations | 1

8. Secondary Outcome: Pharmacists' Use of the Prescription Drug Monitoring Program (PDMP)
Description: Measured at each study visit via an action item checklist to confirm whether the PDMP was inquired to identify the following for each participant: measures of multiple buprenorphine prescriptions, any prescriptions for class II and III medications, and any other information that may be useful for the participant's treatment such as documented drug-related medical interventions or disciplinary charges.
Time Frame: Up to six months
Population: The total number of visits (409) represent the total number of study visits attended in the maintenance phase (n=406) plus early-termination visits (n=3) that are counted separately.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Groups:
- Pharmacist-administered Buprenorphine Maintenance Care: Following buprenorphine/naloxone induction/stabilization with the physician, participants with opioid use disorder will be transferred to the care of pharmacists for the maintenance phase of treatment. Maintenance visits will occur monthly with the pharmacist at the pharmacy location for six months. Buprenorphine/naloxone will be dispensed by the pharmacist at the monthly study visits following participant assessment, communication with the physician, and prescription from the physician.
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
Number analyzed (Participants) | 71
Number analyzed (Visits) | 409
Visits | 396

ADVERSE EVENTS:
Time Frame: 6 months
Description: Collection of safety events was limited to those collected on the Safety Event Response Checklist (SERC-75), which was completed at each visit. There are fifteen types of safety events reported on the SERC-75, including overdoses (ODs), emergency department (ED) visits, hospitalizations, and deaths.
Arm/Group | Pharmacist-administered Buprenorphine Maintenance Care
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 2/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacist-administered Buprenorphine Maintenance Care (N=71)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle cramping from i.v. cocaine use.
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) — 1st, 2nd and 3rd degree burn; resulted in hospitalization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03248947/Prot_SAP_000.pdf